CLINICAL TRIAL: NCT05867342
Title: Effects of Adrenaline Infiltration on Surgical Field of View in Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Hwang, Professor of Otolaryngology - Head & Neck Surgery (OHNS), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40274
Record Dates: First submitted 2018-11-22; First posted 2023-05-22 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Epinephrine; Lidocaine; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Endoscopic sinus surgery (Experimental): Participants receive topical 1:1000 epinephrine plus saline in one nostril, and topical 1:1000 epinephrine plus infiltration of 1% lidocaine with 1:100,000 epinephrine in the other nostril, during endoscopic visualization while undergoing Endoscopic sinus surgery (ESS).
  Interventions: Drug: Epinephrin; Drug: 1% lidocaine with epinephrin 1:100,000; Drug: Saline

INTERVENTIONS:
Drug: Epinephrin — Topical application of 2 pieces of Epinephrin (1:1,000)-soaked cottonoid in nasal cavity
  Other Names: Adrenaline
Drug: 1% lidocaine with epinephrin 1:100,000 — 4 ml intranasal infiltration of 1% lidocaine with epinephrine (1:100,000) at 2 sites (2 ml infiltration at each site)
Drug: Saline — 4 ml intranasal infiltration of saline at 2 sites (2 ml infiltration at each site)

SUMMARY:
In endoscopic sinus surgery a clear surgical field of view is a very important aspect for good surgical outcome. This study is to evaluate the preoperative preparation to acquire best surgical field of view by comparing between the use of topical adrenaline and the use of combination of topical adrenaline with infiltration of 1% lidocaine with adrenaline in patients scheduled for endoscopic sinus surgery for rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with recurrent acute or chronic rhinosinusitis recalcitrant to medical treatment and scheduled for endoscopic sinus surgery

Exclusion Criteria:

* Patients who have asymetrical disease on the two sides (Lund Mackay score difference more than 2)
* Patients who have endoscopic sinus surgery for treatment of tumor or disease other than sinusitis
* Patients with underlying uncontrolled hypertension
* Patients with bleeding disorder or are unable to discontinue antiplatelet or anticoagulant before the surgery
* Patients who are allergic to adrenaline or to xylocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Hwang, MD, Study Director — Stanford University; Navarat Tangbumrungtham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saif AM, Farboud A, Delfosse E, Pope L, Adke M. Assessing the safety and efficacy of drugs used in preparing the nose for diagnostic and therapeutic procedures: a systematic review. Clin Otolaryngol. 2016 Oct;41(5):546-63. doi: 10.1111/coa.12563. Epub 2016 Feb 11. PMID 26452438
- [Background] Yang JJ, Zheng J, Liu HJ, Liu YX, Shen JC, Zhou ZQ. Epinephrine infiltration on nasal field causes significant hemodynamic changes: hypotension episode monitored by impedance-cardiography under general anesthesia. J Pharm Pharm Sci. 2006;9(2):190-7. PMID 16959188
- [Background] Yang JJ, Li WY, Jil Q, Wang ZY, Sun J, Wang QP, Li ZQ, Xu JG. Local anesthesia for functional endoscopic sinus surgery employing small volumes of epinephrine-containing solutions of lidocaine produces profound hypotension. Acta Anaesthesiol Scand. 2005 Nov;49(10):1471-6. doi: 10.1111/j.1399-6576.2005.00869.x. PMID 16223392
- [Background] Moshaver A, Lin D, Pinto R, Witterick IJ. The hemostatic and hemodynamic effects of epinephrine during endoscopic sinus surgery: a randomized clinical trial. Arch Otolaryngol Head Neck Surg. 2009 Oct;135(10):1005-9. doi: 10.1001/archoto.2009.144. PMID 19841339
- [Background] Khosla AJ, Pernas FG, Maeso PA. Meta-analysis and literature review of techniques to achieve hemostasis in endoscopic sinus surgery. Int Forum Allergy Rhinol. 2013 Jun;3(6):482-7. doi: 10.1002/alr.21126. Epub 2012 Dec 16. PMID 23255493
- [Background] Cohen-Kerem R, Brown S, Villasenor LV, Witterick I. Epinephrine/Lidocaine injection vs. saline during endoscopic sinus surgery. Laryngoscope. 2008 Jul;118(7):1275-81. doi: 10.1097/MLG.0b013e31816dd2d9. PMID 18438267
- [Result] Tangbumrungtham N, Hwang PH, Maul X, Borchard NA, Dholakia SS, Patel ZM, Nayak JV, Choby G. The effect of topical epinephrine 1:1000 with and without infiltration of 1% lidocaine with epinephrine 1:100,000 on endoscopic surgical field visualization: a double-blind randomized controlled study. Int Forum Allergy Rhinol. 2020 Feb;10(2):147-152. doi: 10.1002/alr.22468. Epub 2019 Oct 31. PMID 31671251

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: nostrils
Groups:
- 1:1000 Epinephrine Plus Saline; 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine: Participants receive topical 1:1000 epinephrine plus saline in one nostril, and topical 1:1000 epinephrine plus infiltration of 1% lidocaine with 1:100,000 epinephrine in the other nostril, during endoscopic visualization while undergoing Endoscopic sinus surgery (ESS).
Period: Overall Study
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Started | 40; 40 nostrils | 40; 40 nostrils
Completed | 37; 37 nostrils | 37; 37 nostrils
Not Completed | 3; 3 nostrils | 3; 3 nostrils
Not completed — Investigator Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants receive topical 1:1000 epinephrine plus saline in one nostril, and topical 1:1000 epinephrine plus infiltration of 1% lidocaine with 1:100,000 epinephrine in the other nostril.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.46 (16.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Surgical Field Grading Score
Description: The video recording of the endoscopic sinus surgery of the participant was graded by another otolaryngology specialist postoperatively and graded according to Wormald Surgical Field Grading Scale. Scores range from 0 (no bleeding) to 10 (severe bleeding with nasal cavity filling rapidly).
Time Frame: postoperatively (approximately 20 minutes to assess)
Population: Intention-to-treat analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: nostrils
Groups:
- 1:1000 Epinephrine Plus Saline; 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine: Participants receive topical 1:1000 epinephrine plus saline in one nostril, and topical 1:1000 epinephrine plus infiltration of 1% lidocaine with 1:100,000 epinephrine in the other nostril.
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
score on a scale | 3.54 (0.96) | 3.23 (1.14)
Statistical Analysis 1: Comparison: 1:1000 Epinephrine Plus Saline vs 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine; Test type: Other; p = 0.77, t-test, 2 sided — A p-value of < 0.05 would be considered statistically significant

2. Secondary Outcome: Duration of Surgery
Time Frame: intraoperatively (up to 3 hours)
Population: Intention-to-treat analysis set
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: nostrils
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
minutes | 72.05 (35.74) | 54.23 (22.27)
Statistical Analysis 1: Comparison: 1:1000 Epinephrine Plus Saline vs 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine; Test type: Other; p = 0.002, t-test, 2 sided — A p-value of < 0.05 would be considered statistically significant

3. Secondary Outcome: Number of Extra Pledgets Used
Description: A pledget is a small wad of absorbent material used to stop bleeding.
Time Frame: intraoperatively (up to 3 hours)
Population: Intention-to-treat analysis set
Measure: Mean (Standard Deviation); unit: pledgets
Units Other Than Participants: nostrils
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
pledgets | 3.25 (2.82) | 2.63 (3.2)
Statistical Analysis 1: Comparison: 1:1000 Epinephrine Plus Saline vs 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine; Test type: Other; p = 0.126, t-test, 2 sided — A p-value of < 0.05 would be considered statistically significant

4. Secondary Outcome: Estimated Blood Loss During Surgery
Time Frame: intraoperatively (up to 3 hours)
Population: Intention-to-treat analysis set
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: nostrils
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
mL | 95.25 (82.88) | 91.63 (86.98)

5. Secondary Outcome: Postoperative Bloody Discharge Grading Score
Description: Grading of postoperative bloody discharge postoperatively assessed by patient using the 1-week postoperative bleeding questionnaire. Scores range from 0 (no bleeding) to 5 (continuous heavy bleeding necessitating medical care).
Time Frame: 1 week after the surgery (up to 2 minutes to complete assessment)
Population: Intention-to-treat analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: nostrils
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
score on a scale | 2.38 (1.14) | 2.2 (0.213)
Statistical Analysis 1: Comparison: 1:1000 Epinephrine Plus Saline vs 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine; Test type: Other; p = 0.213, t-test, 2 sided — A p-value of < 0.05 would be considered statistically significant

6. Secondary Outcome: Number of Days With Postoperative Bloody Nasal Discharge
Description: Participants indicated number of days with bloody nasal discharge postoperatively using the 1-week postoperative bleeding questionnaire.
Time Frame: 1 week after the surgery (up to 2 minutes to complete assessment)
Population: Intention-to-treat analysis set
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: nostrils
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
days | 2.85 (2.54) | 2.73 (2.35)
Statistical Analysis 1: Comparison: 1:1000 Epinephrine Plus Saline vs 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine; Test type: Other; p = 0.418, t-test, 2 sided — A p-value of < 0.05 would be considered statistically significant

7. Secondary Outcome: Number of Nostrils With Continuous Fresh Bleeding
Description: Number of nostrils with excessive fresh bleeding postoperatively using the 1-week postoperative bleeding questionnaire. Continuous fresh bleeding was defined as bleeding for over 15 minutes.
Time Frame: 1 week after the surgery (up to 2 minutes to complete assessment)
Population: Intention-to-treat analysis set
Measure: Count of Units; unit: nostrils
Units Other Than Participants: nostrils
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
Number analyzed (Participants) | 40 | 40
Number analyzed (nostrils) | 40 | 40
nostrils | 7 | 5
Statistical Analysis 1: Comparison: 1:1000 Epinephrine Plus Saline vs 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine; Test type: Other; p = 0.756, t-test, 2 sided — A p-value of < 0.05 would be considered statistically significant

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 1:1000 Epinephrine Plus Saline | 1:1000 Epinephrine Plus Infiltration of 1% Lidocaine With 1:100,000 Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT05867342/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT05867342/SAP_001.pdf